CLINICAL TRIAL: NCT04423315
Title: Thrombosis Risk Assessment May Predict Clinical Presentation and Length of Hospital Stay in Covid-19 Pneumonia
Brief Title: Thrombosis Risk Assessment and Clinical Presentation of Covid-19 Pneumonia
Acronym: Covid-19
Status: Completed | Type: Observational
Sponsor: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Murat Civan, M.D., Istanbul Nisantasi University
Other Study IDs: 20200504443
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Corona Virus Infection; Thromboembolic Disease
Keywords: covid-19 pneumonia; thromboembolism risk; length of hospitalization
MeSH Terms: conditions — Coronavirus Infections; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with covid-19 pneumonia: patients with covid-19 pneumonia above 18 years old who were diagnosed by pcr testing and computed tomography of thorax

SUMMARY:
Covid-19 mainly affects the respiratory system. Multiple organ dysfunction and a particularly progressive respiratory insufficiency along with a widespread coagulopathy presumed to be due to infection-associated inflammation and the resulting cytokine storm, are strongly associated with high mortality rates. In this study, the association between thrombosis risk and clinical presentation of Covid-19 is investigated.

DETAILED DESCRIPTION:
The severe acute respiratory distress syndrome related coronavirus-2 (SARS-CoV-2) and its clinical presentation as Coronavirus disease 2019 (COVID-19) was first reported in Wuhan, Hubei, China in December 2019. It has spread rapidly from its origin in Wuhan City to other countries of the world over the last several months.

Although it mainly affects the respiratory system , multiple organ dysfunction and a particularly progressive respiratory insufficiency along with a widespread coagulopathy presumed to be due to infection-associated inflammation and the resulting cytokine storm, are strongly associated with high mortality rates. SARS-CoV-2 infection may also lead to thrombotic disease both in the venous and arterial circulation of patients apart from respiratory system due to excessive inflammation, thrombocyte activation, endothelial malfunction, and stasis.

Investigators have reported that both CHADS2 and CHA2DS2-VASc scores were related to mortality in individuals that had stable coronary angina, acute coronary syndrome, Takotsubo syndrome or sick sinus syndrome, apart from atrial fibrillation . In addition, thrombocyte/lymphocyte (PLT/LYM) and neutrophil/lymphocyte (NEU/LYM) ratios on admission were also related with thromboembolic complications in former studies which found them useful to predict prognosis of acute pulmonary embolism, as being one of the thromboembolic complications of Covid-19.

Investigators suggest that the parameters mentioned above should also be studied in terms of thrombotic complications of Covid-19. Thus they aimed to find out potential associations between markers of prothrombotic or inflammatory conditions and some clinical features of Covid-19 pneumonia cases on admission and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with COVID - 19 pneumonia between March 11 th , 2020 and April 25th, 2020 in the emergency, internal medicine and cardiology outpatient clinics.
* patients diagnosed by pcr testing and computed tomography of the chest

Exclusion Criteria:

* patients below 18 years of age
* patients with an alternative aetiology of pneumonia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID - 19 pneumonia diagnosed in the emergency, internal medicine and cardiology outpatient clinics will be included
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | 2 months
  from admission to discharge expressed in days

CONTACTS AND LOCATIONS:
Locations (1):
- Vital Hospital, Bahçelievler, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD excluding names and personal identity numbers will be shared when the research is ready to be submitted for publication

REFERENCES:
- [Background] Wang Q, Ma J, Jiang Z, Ming L. Prognostic value of neutrophil-to-lymphocyte ratio and platelet-to-lymphocyte ratio in acute pulmonary embolism: a systematic review and meta-analysis. Int Angiol. 2018 Feb;37(1):4-11. doi: 10.23736/S0392-9590.17.03848-2. Epub 2017 May 24. PMID 28541022
- [Background] Lippi G, Plebani M. Laboratory abnormalities in patients with COVID-2019 infection. Clin Chem Lab Med. 2020 Jun 25;58(7):1131-1134. doi: 10.1515/cclm-2020-0198. No abstract available. PMID 32119647